CLINICAL TRIAL: NCT00724516
Title: Evaluation Of A Novel Breast Compression Paddle For Wire Localization In Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Caroline Blane, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00013441
Record Dates: First submitted 2008-07-23; First posted 2008-07-29 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Mammography; Biopsy, Needle
Keywords: Mammogram; Biopsy; Needle; Wire; Localization; Compression; Paddle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Novel Breast Compression Paddle (Experimental): Women scheduled to undergo a breast mammography wire localization procedure will have a new breast compression paddle will be used Instead of using the regular wire localization mammography compression paddle.
  Interventions: Device: Novel Breast Compression Paddle

INTERVENTIONS:
Device: Novel Breast Compression Paddle — Instead of using the regular wire localization mammography compression paddle, a new breast compression paddle will be used. The new breast compression paddle is similar to a tennis racquet. It consists of crossing plastic strings that are strung tightly in a frame. The needle/wire can be inserted anywhere between the strings.

SUMMARY:
The purpose of this study is to evaluate the functionality of a new breast compression paddle used in mammography for wire localization.

DETAILED DESCRIPTION:
Presently, the breast compression paddles that are used in mammography for wire localization are made of plastic and contain a relatively small rectangular shaped opening through which the wire is placed in the breast. When technologists use this paddle, they must carefully position the breast such that the rectangular opening is above the region for wire localization. A novel paddle has been developed which increases the wire localization access area tremendously and should therefore make it easier to perform the procedure. The purpose of this study is to evaluate the functionality of this new compression paddle. The new compression paddle was developed by Biomedical Engineering students in conjunction with Radiologists and a Medical Physicist at the University of Michigan. It was designed and manufactured for a student project in the Mechanical Engineering 450/599 course at the University of Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Women who are scheduled to undergo a wire localization procedure on the digital mammography unit at the University of Michigan Cancer Center

Exclusion Criteria:

* Men
* Pregnant Women
* Lactating Women
* Prisoners
* Children under the age of 18
* Mentally impaired individuals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the newly designed breast compression paddle. | 1 year
  To objectively determine if the functionality of this new breast compression paddle allows for easier access to the breast during wire localization.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Blane, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No